CLINICAL TRIAL: NCT01537965
Title: Evaluation of Innovative Ultrasonic Techniques for Non-invasive Diagnosis of Liver Fibrosis in Patients With Chronic Viral Hepatitis B or C
Acronym: FIBRECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Clinical Investigation Centre for Innovative Technology Network (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DCIC 11 03
Record Dates: First submitted 2011-12-15; First posted 2012-02-23 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Liver Fibrosis
Keywords: hepatitis; fibrosis; elastography
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Fibroscan® of Echosens, Aixplorer® of Supersonic Imagine, Aplio XG of Toshiba, QRS software developed by Pr I.Bricault, Acuson S2000 of Siemens — Five ultrasounds exams are realised:
  * elastography with Fibroscan®
  * ultrasound elastography in supersonic mode with Aixplorer®
  * ultrasound analysis of the surface liver with QRS software,
  * quantification of acoustic structure with Aplio XG,
  * elastography ARFI with Acuson S2000.

SUMMARY:
The non-invasive assessment of liver fibrosis in chronic viral hepatitis B and C is now entering clinical practice. It is based on blood tests, especially FibroMetre® and Fibrotest® and on elastography with the Fibroscan®. Despite the overall satisfactory diagnostic performance for all of these tests (AUROC ranging from 0.80 to 0.90 depending on the study) for the discrimination of F≤1 versus F≥2, the positive and negative predictive values , however, are far from be perfect in a given patient. With these technique, failures are also possible and the measures do not meet quality standards that increase the risk of misclassification. It would be particularly useful to have new generation techniques with a better diagnostic performance.

In this project, in response to the problems presented above, we propose to evaluate the diagnostic performance of five innovative ultrasonic techniques for the non-invasive diagnosis of fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* patient with an Ac-HCV positive and RNA HCV positive or AgHBs-positive,
* naive to treatment or not receiving treatment for viral eradication in six months,
* patient for whom a liver biopsy size less than 15 mm, regardless of the number of portal tracts present or fragments, is being considered or has been performed between two and one month before inclusion,
* Patient affiliated to social security or similar regime,
* patients who signed consent for participation in the study.

Exclusion Criteria:

* patient with anti-HIV Ac positive (latter result not older than 12 months and in the absence of risk factors)
* chronic liver disease due to other causes than HCV (hemochromatosis, autoimmune hepatitis, autoimmune disease, metabolic liver disease, alcoholic liver disease, alcoholic liver disease, exposure to toxins ...)
* chronic alcohol consumption >30g/day in men and >20g/day in women
* history of severe systemic disease,
* HCV treatment with anti-viral or anti-fibrotic referred to within the last 6 months,
* immunosuppressive therapy: corticosteroids, Imurel, cyclosporine, tacrolimus, Cellcep,
* patient with an active implantable medical device,
* protected person referred to in Articles L1121-5 to L1121-8 of the Code of Public Health

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
In patients with chronic viral hepatitis B or C, evaluate the performance for the diagnosis of significant fibrosis (F≤1 versus F≥2) of elastography in mode supersonic compared with elastography (FibroScan®), the gold standard liver biopsy. | two years
  Comparison 2-2 of areas under the ROC curve obtained for the different modalities (Fibroscan® vs Aixplorer®).

SECONDARY OUTCOMES:
Compare the performance for the diagnosis of significant fibrosis of the liver contours regularity quantification and of the homogeneity of the hepatic parenchyma, and biological tests of fibrosis, the gold standard is liver biopsy. | two years
  Comparison 2-2 of areas under the ROC curve obtained for the different modalities (Fibrotest®, Fibromètre®, Acoustic Structure Quantification, Quantification of the Surface Regularity, elastography ARFI)
Evaluate the diagnostic performance of each technique (ultrasound innovative and organic) for severe fibrosis (F<3 vs F≥3) and cirrhosis (F<4 vs F≥4). | two years
  Comparison 2-2 of areas under the ROC curve obtained for the different modalities (Fibrotest®, Fibromètre®, elastography with Fibroscan®, elastography in mode supersonic, Acoustic Structure Quantification, Quantification of the Surface Regularity, elastography ARFI)
Evaluate the diagnostic performance of all approaches to all stages of fibrosis took 2 by 2 (F1 vs. F2, F2 vs. F3, F3 vs. F4) | two years
  Comparison 2-2 of areas under the ROC curve obtained for the different modalities (Fibrotest®, Fibromètre®, elastography with Fibroscan®, elastography in mode supersonic, Acoustic Structure Quantification, Quantification of the Surface Regularity, elastography ARFI)
Evaluate the performance of the main diagnostic modalities chosen from previous results in the two sub-populations: patients with hepatitis B and those with hepatitis C | two years
  Comparison of areas under the ROC curve obtained in the two sub-population (hepatisis B and C) for the main diagnostic modalities chosen from previous results.
Kappa intra-observer coefficient of ultrasonic techniques | two years
Propose, based on previous results, a hierarchical strategy for using these innovative ultrasonic techniques used in combination with Fibroscan ® and the biological tests currently available (Fibrotest ®, FibroMetre ®). | two years
  proportion of patients correctly classified by the new strategy for each grade of fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Leroy, Pr, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble, France